CLINICAL TRIAL: NCT03943693
Title: Dual Shock Versus Single Shock Synchronized External Direct Current Cardioversion for Atrial Fibrillation - A Double-blinded Randomized Trial
Brief Title: Dual Versus Single Shock for Cardioversion of Atrial Fibrillation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10276
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Atrial Fibrillation
Keywords: Cardioversion
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Single Shock Group (Active Comparator): Patients randomized to single shock will then be treated initially with a 200 Joule shock through the antero-posterior pads only.
  Interventions: Device: Single shock
- Double Shock Group (Active Comparator): Patients randomized to the dual shock group will have two near-simultaneous 200-Joule shocks delivered through the two sets of pads (antero-posterior position and right infraclavicular-axillary position). The first of these shocks will be synchronized.
  Interventions: Device: Double shock

INTERVENTIONS:
Device: Double shock — Patients randomized to the dual shock group will have two near-simultaneous 200-Joule shocks delivered through the two sets of pads (antero-posterior position and right infraclavicular-axillary position). The first of these shocks will be synchronized. If the first attempt with this approach fails to terminate atrial fibrillation a second attempt will be made using the same approach. If the second attempt fails the dual shock approach will be considered to have failed and further treatment will be determined by the primary team/attending cardiologist.
  Arms: Double Shock Group
Device: Single shock — Patients randomized to single shock will then be treated initially with a 200 Joule shock through the antero-posterior pads only. A repeat attempt will be made using the same approach if the initial shock fails. If the second attempt fails, the single shock approach will be considered to have failed. Patients will be crossed over to dual shock therapy while under the same sedation episode. For cross-over patients, two near-simultaneous 200-Joule shocks will be delivered through the two sets of pads already in position. If this fails further treatment will be determined by the primary team/attending cardiologist.
  Arms: Single Shock Group

SUMMARY:
The investigators aim to investigate the immediate success rate (rate of termination of atrial fibrillation) of dual shock cardioversion compared with standard single shock cardioversion in patients with baseline characteristics adversely influencing successful cardioversion. Baseline characteristics known to reduce the success rate of single shock cardioversion include: increased body mass index (BMI), chronic obstructive pulmonary disease, sleep apnea, enlarged left atrium, longer duration of atrial fibrillation and use of amiodarone.

DETAILED DESCRIPTION:
Patient Enrollment Patient enrollment will be open enrollment to inpatient/outpatients who meet the inclusion/exclusion criteria listed above. This is a double-blinded study with randomization to dual shock or standard single shock synchronized cardioversion for patients requiring cardioversion for atrial fibrillation. Randomization will be performed using a standard computer-based randomization system.

Cardioversion will be performed with Zoll R series Defibrillator, which was approved by the FDA in 2017 for use as a defibrillator, with a 510K approval for use in cardioversion of atrial arrhythmias. After obtaining consent, before sedation is administered, all patients will have 2 pads placed in the antero-posterior pad position on the left chest (guideline recommended position for cardioversion of atrial fibrillation) and an additional 2 pads placed in the standard Ventricular Tachycardia/Advanced Cardiac Life Support positions, where the anterior pad is centered over the right infraclavicular space and the apical pad is placed over the left axilla . All patients will be sedated using propofol administered by anesthesiology or a combination of fentanyl and midazolam administered by cardiology staff.

Patients randomized to single shock will then be treated initially with a 200 Joule shock through the antero-posterior pads only. A repeat attempt will be made using the same approach if the initial shock fails. If the second attempt fails, the single shock approach will be considered to have failed. Patients will be crossed over to dual shock therapy while under the same sedation episode. For cross-over patients, two near-simultaneous 200-Joule shocks will be delivered through the two sets of pads already in position. If this fails further treatment will be determined by the primary team/attending cardiologist.

Patients randomized to the dual shock group will have two near-simultaneous 200-Joule shocks delivered through the two sets of pads (antero-posterior position and right infraclavicular-axillary position). The first of these shocks will be synchronized. If the first attempt with this approach fails to terminate atrial fibrillation a second attempt will be made using the same approach. If the second attempt fails the dual shock approach will be considered to have failed and further treatment will be determined by the primary team/attending cardiologist.

Primary Endpoint - Successful termination of atrial fibrillation after initial Direct Current Ccardioversion (DCCV). Successful cardioversion = immediate termination of atrial fibrillation with electrocardiographic (ECG) evidence of atrial fibrillation (AF) termination. The physician deciding whether AF was successfully terminated will be blinded to whether the shock was with single or dual shocks. - Partial success will be considered if atrial fibrillation is terminated by the second attempt using the same approach. Secondary Endpoints - Maintenance of normal sinus rhythm at one hour post cardioversion - Presence of symptomatic skin burn (symptoms rated on a scale of 1-10) - Thromboembolic complications - Ventricular Arrhythmias requiring additional shock therapy Documentation of Anticoagulation All patients need to have established therapeutic anticoagulation. Either 1) Therapeutic warfarin (with International normalized ratio (INR) >2) or therapeutic doses of apixaban, dabigatran, rivaroxaban or edoxaban for at least 3 consecutive weeks before and with plans to continue 4 weeks after cardioversion. 2) Therapeutic anticoagulation with intravenous heparin or therapeutic subcutaneous enoxaparin or non-vitamin K oral anticoagulant if atrial fibrillation episode is known to be of recent onset (<48 hours), with anticoagulation to continue for at least one week post cardioversion. 3) Sub-therapeutic or no anticoagulation preceding cardioversion, but transesophageal echocardiogram (TEE) confirming absence of intra-cardiac thrombus. Therapeutic anticoagulation should be administered just prior to cardioversion and planned to continue for at least 4 weeks post cardioversion.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient or inpatients with atrial fibrillation sent for elective direct current cardioversion (DCCV) with at least 1 of the following risk factors will be included:

  * BMI >30
  * History of Chronic Obstructive Pulmonary Disease/emphysema/asthma
  * Significant Valvular heart disease (at least moderate regurgitation/stenosis)
  * History of Heart Failure with preserved Ejection Fraction/Heart Failure with reduced Ejection Fraction
  * Cardiomyopathy with ejection fraction <40%
  * Left atrium anterior-posterio (AP) dimension >4.5cm
  * Presence of Left ventricular hypertrophy (≥1.1cm septal/posterior wall M-mode) on transthoracic echocardiogram
  * History of sleep apnea

Exclusion Criteria:

* Consent not obtained
* <18 y.o.
* >80 y.o.
* Not adequately anti-coagulated
* Patient hemodynamically unstable and DCCV required as an emergent procedure
* Prisoners or pregnant patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Cardioversion to sinus rhythm | Immediately following cardioversion
  Successful termination of atrial fibrillation after initial DCCV. Successful = cardioversion = immediate termination of atrial fibrillation

SECONDARY OUTCOMES:
Maintenance of normal sinus rhythm at one hour post cardioversion | Within 24 hours
Presence of symptomatic skin burn | Immediately following cardioversion
  Symptoms rated on a scale 1-10
Thromboembolic complications | Within 24 hours
Ventricular arrhythmias requiring additional shock therapy | Immediately following cardioversion

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Lockwood, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Science Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saliba W, Juratli N, Chung MK, Niebauer MJ, Erdogan O, Trohman R, Wilkoff BL, Augostini R, Mowrey KA, Nadzam GR, Tchou PJ. Higher energy synchronized external direct current cardioversion for refractory atrial fibrillation. J Am Coll Cardiol. 1999 Dec;34(7):2031-4. doi: 10.1016/s0735-1097(99)00463-5. PMID 10588220
- [Result] Chugh SS, Havmoeller R, Narayanan K, Singh D, Rienstra M, Benjamin EJ, Gillum RF, Kim YH, McAnulty JH Jr, Zheng ZJ, Forouzanfar MH, Naghavi M, Mensah GA, Ezzati M, Murray CJ. Worldwide epidemiology of atrial fibrillation: a Global Burden of Disease 2010 Study. Circulation. 2014 Feb 25;129(8):837-47. doi: 10.1161/CIRCULATIONAHA.113.005119. Epub 2013 Dec 17. PMID 24345399
- [Result] Boriani G, Diemberger I, Biffi M, Domenichini G, Martignani C, Valzania C, Branzi A. Electrical cardioversion for persistent atrial fibrillation or atrial flutter in clinical practice: predictors of long-term outcome. Int J Clin Pract. 2007 May;61(5):748-56. doi: 10.1111/j.1742-1241.2007.01298.x. PMID 17493088
- [Result] Larsen MT, Lyngborg K, Pedersen F, Corell P. [Predictive factors of maintenance of sinus rhythm after direct current (DC) cardioversion of atrial fibrillation/atrial flutter]. Ugeskr Laeger. 2005 Sep 5;167(36):3408-12. Danish. PMID 16159494
- [Result] Vinolas X, Freire F, Romero-Menor C, Alegret JM. [Predictors of reversion to sinus rhythm previous to electrical cardioversion in patients with persistent atrial fibrillation treated with anti-arrhythmic drugs]. Med Clin (Barc). 2013 Apr 20;140(8):351-5. doi: 10.1016/j.medcli.2012.02.026. Epub 2012 Sep 14. Spanish. PMID 22982132
- [Result] Marrouche NF, Bardy GH, Frielitz HJ, Gunther J, Brachmann J. Quadruple pads approach for external cardioversion of atrial fibrillation. Pacing Clin Electrophysiol. 2001 Sep;24(9 Pt 1):1321-4. doi: 10.1046/j.1460-9592.2001.01321.x. PMID 11584453